CLINICAL TRIAL: NCT02874664
Title: An Intensive QT/QTc Study to Investigate the Effects of Rovalpituzumab Tesirine on Cardiac Ventricular Repolarization in Subjects With Small Cell Lung Cancer
Brief Title: A Study of Rovalpituzumab Tesirine to Study Cardiac Ventricular Repolarization in Subjects With Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stemcentrx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRX001-007
Record Dates: First submitted 2016-08-16; First posted 2016-08-22 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — rovalpituzumab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rovalpituzumab Tesirine (Experimental): 0.3 mg/kg rovalpituzumab tesirine intravenously on Day 1 of every 6-week treatment cycle for 2 cycles omitting every third cycle
  Interventions: Drug: Rovalpituzumab Tesirine

INTERVENTIONS:
Drug: Rovalpituzumab Tesirine — Rovalpituzumab tesirine is a DLL3 targeted antibody drug conjugate (ADC)
  Other Names: SC16LD6.5

SUMMARY:
Study to evaluate the effect of rovalpituzumab tesirine on cardiac ventricular repolarization in subjects with small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive-stage small-cell lung cancer (SCLC).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate hematologic and organ function as confirmed by laboratory values

Exclusion Criteria:

* Clinically significant cardiac abnormalities including QRS duration of >120 msec; QTcF >470 msec for women and >450 msec for men; Abnormal cardiac rhythm; Clinically significant cardiac valve abnormality; Documented history of left ventricular ejection fraction <0.30 within 6 months; Permanent pacemaker or automatic implantable cardioverter defibrillator; History of torsades de pointes, congenital long QT syndrome, or family history of long QT syndrome or sudden death
* Recent or ongoing serious infection
* Women who are pregnant or breastfeeding
* Prior exposure to a pyrrolobenzodiazepine (PBD)-based drug, prior participation in a rovalpituzumab tesirine clinical trial, or known hypersensitivity to rovalpituzumab tesirine or excipient contained in the drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Change in QTcF interval from baseline QTcF following treatment with rovalpituzumab teserine as measured by extracting quantitative ECG parameters from ambulatory Holter monitors. | 12 weeks

SECONDARY OUTCOMES:
Change in RR interval from baseline RR following treatment with rovalpituzumab teserine as measured by extracting quantitative ECG parameters from ambulatory Holter monitors. | 12 weeks
Change in PR interval from baseline PR following treatment with rovalpituzumab teserine as measured by extracting quantitative ECG parameters from ambulatory Holter monitors. | 12 weeks
Change in QRS duration interval from baseline QRS duration following treatment with rovalpituzumab teserine as measured by extracting quantitative ECG parameters from ambulatory Holter monitors. | 12 weeks
Change in waveform composition interval from baseline waveform composition following treatment with rovalpituzumab teserine as measured by extracting quantitative ECG parameters from ambulatory Holter monitors. | 12 weeks
Relationship between plasma rovalpituzumab tesirine concentration and change in QTcF interval from baseline. | 12 weeks
Incidence of proarrhythmic adverse events stratified by change in QTcF from baseline of less than 10 ms or greater than 10 ms. | 12 weeks
Incidence of adverse events. | From first dose through 30 days post-last-dose
Objective response rate | Baseline, every 6 weeks until 6 months, then every 12 weeks until disease progression, assessed up to 24 months.
Duration of response | Baseline, every 6 weeks until 6 months, then every 12 weeks until disease progression, assessed up to 24 months.
Progression free survival | Baseline, every 6 weeks until 6 months, then every 12 weeks until disease progression, assessed up to 24 months.
Overall survival | Baseline, every 6 weeks until 6 months, then every 12 weeks until disease progression, assessed up to 24 months.
Clinical benefit ratio | Baseline, every 6 weeks until 6 months, then every 12 weeks until disease progression, assessed up to 24 months.
Maximum Plasma Concentration (Cmax) | Cycles 1 and 2: Day 1 (predose, 30 min, 2 and 4 hours postdose) and days 2,3,4,8,15,and 29; Cycles 4,5,7,8: Day 1 predose and 30 min postdose.
Area Under the Curve (AUC) | Cycles 1 and 2: Day 1 (predose, 30 min, 2 and 4 hours postdose) and days 2,3,4,8,15,and 29; Cycles 4,5,7,8: Day 1 predose and 30 min postdose.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Da Costa, PharmD, Study Director — AbbVie
Locations (15):
- United States (13):
  - University of California Los Angeles, Los Angeles, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital-Cancer Centre, Ottawa, Ontario